CLINICAL TRIAL: NCT05991739
Title: Pilot Testing of a Structural Racism Intervention for Immigrant Latinx Families: Blending of Implementation Science and Community-Engaged Research
Brief Title: Pilot Testing of a Structural Racism Intervention for Immigrant Latinx Families
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: The Resurrection Project (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-0108; CTSA UL1TR002003 (Other Grant/Funding Number: UIC Center for Clinical and Translational Science)
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Stress, Psychological; Mental Health Wellness
Keywords: immigrant families; stress intervention; structural racism; latino
MeSH Terms: conditions — Stress, Psychological; Systemic Racism

STUDY DESIGN:
Intervention Model Description: This study will randomize 35 parent-youth dyads to the treatment arm or waitlist-control arm using block randomization. Each group will have 7-9 dyads, with two groups running simultaneously (treatment arm) and the remaining two groups running in three months (waitlist-control arm). After all participants are enrolled, families will be randomly selected to participate in either the treatment arm (immediate start) or waitlist-control arm (delayed start after 3 months).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Participants in the treatment arm will begin the FIESTA intervention immediately (Time 1).
  Interventions: Behavioral: Familias Inmigrantes Empoderándose contra eStrés Tomando Acción (FIESTA)
- Waitlist-Control (Other): Participants in the waitlist-control arm will wait approximately three months for the FIESTA intervention (Time 2).
  Interventions: Behavioral: Familias Inmigrantes Empoderándose contra eStrés Tomando Acción (FIESTA)

INTERVENTIONS:
Behavioral: Familias Inmigrantes Empoderándose contra eStrés Tomando Acción (FIESTA) — FIESTA is a 10-session, group intervention led by community health workers that offers strategies related to individual stress management, family coping and communication, and community navigation.

SUMMARY:
The purpose of this study is to evaluate a new, community-based, group intervention called FIESTA (Familias Inmigrantes Empoderándose contra eStrés Tomando Acción) to understand how well it helps Latinx immigrant families deal with the impact of stress due to structural racism. Structural racism is defined as the policies, practices, and norms that work together to limit equal opportunities for minority communities. For Latinx immigrant families, this can include fears of deportation, lack of bilingual providers, and discrimination. These experiences of structural racism can turn into stress, which impacts well-being and mental health.

Researchers will investigate if: 1) FIESTA lowers stress and mental health symptoms (anxiety/depression) and increases feelings of empowerment, improved knowledge of resources, better parent-youth relationship quality, and higher use of healthy coping skills; and 2) FIESTA is feasible (easy to carry out), acceptable (agreeable or satisfactory), and appropriate (relevant to the needs of Latinx families).

FIESTA is ten-sessions and will be led by two community health workers. Researchers will enroll 35 parent-adolescent dyads (35 study-eligible parents and 35 study-eligible youth) in the initial study. This study will randomize parent-youth dyads to the treatment arm or waitlist-control arm using block randomization. In other words, participants will be randomly assigned to one of two groups, the First Group, or the Second Group. The First Group will begin immediately, and the Second Group will begin after three months. Data will be collected at baseline and three- and six-month post-baseline.

DETAILED DESCRIPTION:
The aim of the study is to pilot test a new, evidence-informed group intervention (FIESTA) among Latina immigrant mothers and youth (ages 14-17) and determine preliminary evidence as well as acceptability, appropriateness, and feasibility. FIESTA was developed in collaboration with a local community-based organization, the research team's established community partner.

Participants will be recruited through the research team's established community partnership. To participate in FIESTA, both the caregiver and child are required to participate. Researchers will enroll 35 parent-adolescent dyads (35 study-eligible parents and 35 study-eligible youth) in the initial pilot study. This study will randomize parent-youth dyads to the treatment arm or waitlist-control arm using block randomization. Each group will have 7-9 dyads, with two groups running simultaneously (treatment arm) and the remaining two groups running in three months (waitlist-control arm). After all participants are enrolled, families will be randomly selected to participate in either the treatment arm (immediate start) or waitlist-control arm (delayed start after 3 months). Participants in the treatment arm will begin the intervention immediately (Time 1) and the waitlist-control arm will wait approximately three months for the intervention (Time 2). All participants will be reassessed at Time 2 (after 3-months) and again at Time 3 (after 6-months), once the wait-control group has completed the intervention. After the intervention (Time 2 for the treatment arm and Time 3 for the waitlist-control arm), participants will be asked a series of questions about the FIESTA intervention to assess for appropriateness, acceptability, and feasibility. All data collection will be completed by the research team.

Each FIESTA group will be led by two community health workers who will not be involved in the research and will not know who participates in the study. The community health workers will meet the following criteria: 1) have participated in a leadership role at the community-based organization or an affiliated organization for at least one year; 2) have experience facilitating at least one workshop; and 3) attend and participate in a three-day training for FIESTA led by the PI.

Each FIESTA session is two hours and will occur over ten weeks. FIESTA covers strategies related to individual stress management, family coping and communication, and community navigation. Throughout the sessions, there is an emphasis on sharing community-based resources if parents or youth are interested in obtaining future services. Each session will run parent and youth groups simultaneously, with a parent-youth activity built into each session. Parent and youth groups will be delivered separately to allow for a private space to discuss sensitive topics and practice skills. Material delivered to youth has been developmentally tailored. Session One provides participants with psychoeducation of stress, including the behavioral, emotional, and cognitive signs of stress, and focuses on recognizing stressors within Latinx communities. Session Two focuses on introducing the cognitive triangle and encourages participants to identify how their feelings, thoughts, and behaviors are connected. Participants will also learn evidence-based relaxation and mindfulness techniques that they will practice throughout the remainder of the sessions. Session Three teaches challenging negative thoughts and problem-solving techniques, using vignettes geared towards Latinx families (e.g., navigating language constraints at work). Session Four focuses on improving communication between parents and their children by teaching "I statements" and active listening through a series of role plays. Session Five is facilitated by an outside consultant recommended by the community partner and teaches about empowerment, the relationship between empowerment and self-esteem, and recognition of internal strengths and external support systems. Session Six focuses on principles developed from Know Your Rights trainings, including understanding rights when interacting with ICE and police and how to create a family emergency plan. Session Seven encourages participants to share their stress related to the Latinx experience, providing a safe space for participants to process their stress and collectively practice stress management skills learned in previous sessions. Session Eight aims to teach participants about advocacy, particularly advocacy in schools, and provides school- and community-based resources meant to help families navigate the school system. Session Nine focuses on financial wellness among immigrant communities, including creating budgets and learning about financial resources, including lending circles and financial aid. Session Ten is the culmination of FIESTA and allows participants to share their successes with the group, review skills, and discuss any linkages to resources. After Session 10, FIESTA will host a celebration where friends and family have a chance to share in the successes of participants.

ELIGIBILITY:
Inclusion Criteria:

Caregiver/Parent

* Identification as a Latina immigrant woman over the age of 18 years old
* Parent or primary caregiver of a youth between the ages of 14-17

Youth

* Identification as a Latinx adolescent between the ages of 14-17
* Child of a primary caregiver (mother) who identifies as a Latina immigrant

Exclusion Criteria:

* Adults and youth unable to cognitively participate in the group or adults who are unable to consent

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Hispanic Stress Inventory 2 | Baseline, 3 months, and 6 months
  Self-reported (parent and youth) stress due to structural racism
Perceived Stress Scale | Baseline, 3 months, and 6 months
  Self reported (parent and youth) daily stress
Parent-Reported Outcome Measurement Information System Depression and Anxiety Short Form | Baseline, 3 months, and 6 months
  Self reported (parent and youth) depression and anxiety symptoms

SECONDARY OUTCOMES:
Brief Coping Orientation to Problems Experienced Inventory | Baseline, 3 months, and 6 months
  Self reported (parent and youth) individual coping
Family Crisis Oriented Personal Evaluation Scales | Baseline, 3 months, and 6 months
  Self reported (parent and youth) family coping
Parent-Adolescent Communication Scale | Baseline, 3 months, and 6 months
  Self reported (parent and youth) parent-child relationship quality
General Self-Efficacy Scale | Baseline, 3 months, and 6 months
  Self reported (parent and youth) empowerment
Knowledge of Resources | Baseline, 3 months, and 6 months
  Self reported (parent and youth) knowledge of resources in the community

OTHER OUTCOMES:
Implementation Interview | Post-intervention (Time 2 for the treatment arm and Time 3 for the waitlist-control arm)
  Self reported (parent and youth); a series of interview questions will be asked to assess the appropriateness, acceptability, and feasibility of FIESTA

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie A Torres, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No